CLINICAL TRIAL: NCT06553612
Title: Impact of a Multidisciplinary Assessment in Day Hospitalization Versus Standard Care on the Deployment of Supportive Oncology Care Recommended by the Personalized Post-cancer Plan in Patients at the End of Initial Treatment for Gynecological Ovarian and Endometrial Cancer Endometrial Cancer
Acronym: AFTERGYN2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A02554-41
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Gynecologic Cancer; Remission
Keywords: supportive oncology care; personalized post-cancer plan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Delivery of personalized post-cancer plan with multidisciplinary assessment of oncology support care needs in a day hospital
  Interventions: Other: Multidisciplinary assessment
- Control group (Active Comparator): Delivery of a personalized post-cancer plan without a day hospital
  Interventions: Other: Standard assesment
- Cohort (Other): Follow-up as part of an observational cohort
  Interventions: Other: Observational cohort

INTERVENTIONS:
Other: Multidisciplinary assessment — Delivery of a personalized post-cancer plan with multidisciplinary assessment of oncology support care needs in a day hospital
  Arms: Experimental group
Other: Standard assesment — Delivery of a personalized post-cancer plan without a day hospital
  Arms: Control group
Other: Observational cohort — Patients with no cancer sequelae, no adverse effects and no need for oncological support care will not be randomized, but will be followed as part of an observational cohort
  Arms: Cohort

SUMMARY:
This project proposes a structuring of supportive oncology care for the recovery phase after gynecological cancer (ovarian/trope/peritoneum or endometrium). Patients will be divided into three groups based on the identification of oncological support care needs. Patients with supportive oncology care needs will be randomized into two groups: the experimental group, receiving a personalized post-cancer plan with a multidisciplinary assessment of supportive oncology care needs in a day hospital and coordinated follow-up by the referring study nurse, and the control group, receiving a personalized post-cancer plan without a day hospital. Randomization will be stratified according to tumor location (ovary vs. endometrium), use of supportive oncology care during treatment, and treatment center. Patients with no need for supportive oncology care will be followed in an observational cohort. The main objective is to identify and manage the supportive oncology care needs of patients in remission from endometrial or ovarian cancer to improve their quality of life and post-treatment follow-up. A medico-economic analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years
* Patients in remission from first-line treatment of endometrial or ovarian/tumor/peritoneal cancer.
* Patient who has completed her initial treatment; patients on maintenance therapy are eligible.
* Fluency in French
* Patient with access to a telephone line
* Patient affiliated to a social security scheme
* Signature of informed consent prior to any specific study procedure

Exclusion Criteria:

* Any associated medical or psychiatric condition that could compromise the patient's ability to participate in the study
* Patient with locoregional or metastatic recurrence
* Patient deprived of liberty, under guardianship or curatorship
* Simultaneous participation in a therapeutic clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2027-09-07 (Estimated); Study Completion 2028-06-07 (Estimated)

PRIMARY OUTCOMES:
Compare the proportion of patients for whom the supportive oncology care recommended in the personalized post-cancer plan has been implemented. | 6 months after delivery of personalized post-cancer plan, i.e. about 8 months after inclusion
  The primary criterion is the proportion of patients who have implemented at least one of the supportive oncology treatments recommended in the personalized post-cancer plan within 6 months of receiving the personalized post-cancer plan.

SECONDARY OUTCOMES:
Comparison, 12 months after delivery of the personalized post-cancer plan, of the impact of the intervention on the improvement of side effects and/or sequelae identified at the end of the initial treatments. | 12 months after delivery of personalized post-cancer plan, i.e. about 14 months after inclusion
  Proportion of patients presenting, at 12 months, an improvement (reduction in grade according to CTCAE v5.0 criteria) in at least one of the side effects and/or sequelae identified at the end of the initial treatments according to the INCa identification grids (1st and 2nd levels).

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU, Besançon, Besançon
  - François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - Hopital Diaconesses Croix Saint-Simon, Paris
  - Hopital Europeen George Pompidou, Paris
  - Hôpital COCHIN, Paris
  - Institut Curie, Paris
  - Hopital privé des Côtes d'Armor, Plérin
  - Institut Curie, St Cloud, Saint-Cloud
  - CHU, Saint Etienne, Saint-Etienne
  - CHU, Strasbourg
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No